CLINICAL TRIAL: NCT06703372
Title: Effectiveness Of Photobiomodulation In Treatment Of Xerostomia In Type Ii Diabetic Patients (A Randomized, Controlled Clinical Trial)
Brief Title: Photobiomodulation In Treatment Of Xerostomia In Type Ii Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0404-9/22
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Xerostomia; Diabetes Mellitus
MeSH Terms: conditions — Xerostomia; Diabetes Mellitus | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode laser (Experimental)
  Interventions: Other: Diode Laser 980 nm, 0.2W
- placebo diode laser (Placebo Comparator)
  Interventions: Other: Placebo Diode laser

INTERVENTIONS:
Other: Diode Laser 980 nm, 0.2W — diode laser will be used at an operating wavelength of 980 nm, with adoption of the due safety measures in all cases. Laser irradiation will be applied bilaterally to the skin over the area of the submandibular and parotid glands. Irradiation will be applied externally to the parotid gland on a continuous basis and likewise to the submandibular gland moving the laser very slowly over the gland zone
  Arms: Diode laser
Other: Placebo Diode laser — the tip of the instrument will be sealed with blue rubber to prevent the passage of light
  Arms: placebo diode laser

SUMMARY:
Xerostomia is a major oral health problem that if not recognized and treated can have a significant effect on a patient's quality of life. It leads to difficulties with speech, swallowing and taste alteration. Pathological causes of xerostomia are divided into local and systemic factors. Local factors include smoking, salivary gland diseases and head and neck radiation therapy. Systemic factors include autoimmune diseases as Sjögren syndrome and hormonal disorders as Diabetes Mellitus. Photobiomodulation (PBM) previously known as Low Level Laser Therapy (LLLT) is the application of red and near infra-red light over injuries or lesions to improve wound and soft tissue healing, reduce inflammation and give relief for both acute and chronic pain. It also has grabbed the attention over the last few years as an effective treatment for xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus suffering from xerostomia and on oral hypoglycemic drugs.
* Glycated hemoglobin less than 7%.
* Duration of diabetes mellitus not less than 4 years and not more than 8 years

Exclusion Criteria:

* Patients receiving any drugs that cause hyposalivation.
* Patients with any systemic disease reported to produce hyposalivation (sjogren's syndrome, hepatitis c, rheumatoid arthritis and lupus erythematosus).
* Patients receiving chemotherapy and radiotherapy.
* Individuals with skin lesions in the treatment zone to avoid any complications occurring in this area by laser exposure

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in severity of xerostomia | baseline, 2 weeks, 4 weeks, 6 weeks and 12 weeks
  Summated Xerostomia Inventory-Dutch Version questionnaire (SXI-D) version will be used to assess the severity of xerostomia.
  Questions:
  * My mouth feels dry when eating a meal.
  * My mouth feels dry.
  * I have difficulty in eating dry foods.
  * I have difficulties swallowing certain foods.
  * My lips feel dry
  Scores:
  * Never scoring 1
  * Occasionally scoring 2
  * Ever scoring 3
Change in unstimulated salivary flow rate | baseline, 2 weeks, 4 weeks, 6 weeks and 12 weeks
  Hypo-salivation will be determined if the unstimulated salivary flow rate is 0.1- 0.2 ml/min or less
Change in stimulated salivary flow rate | baseline, 2 weeks, 4 weeks, 6 weeks and 12 weeks
  Whole-mouth SFR measurement will be conducted at every follow-up time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt